CLINICAL TRIAL: NCT01959867
Title: Clinical Study Comparing Two-Stage Breast Reconstruction Following Mastectomy With and Without the Use of SurgiMend® PRS Fetal Bovine Collagen Matrix in Patients With Pre-Mastectomy Radiation Therapy
Brief Title: SurgiMend in Two-stage Implant-based Breast Reconstruction in Patients With Pre-Mastectomy Radiotherapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEI-BR-001
Record Dates: First submitted 2013-09-27; First posted 2013-10-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: mastectomy; breast reconstruction; bovine; ADM; breast cancer; breast implants; breast expanders; radiation therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SurgiMend® PRS (ADM) (Experimental): Subjects enrolled in to this cohort will receive SurgiMend® PRS (ADM) product during the first stage of the reconstruction (expander insertion).
  Interventions: Device: SurgiMend® PRS
- No Intervention (Other): Subjects enrolled in to this cohort will not receive an acellular dermal matrix (ADM) product during the first stage of the reconstruction (expander insertion).
  Interventions: Other: No Intervention

INTERVENTIONS:
Device: SurgiMend® PRS — Subjects enrolled in to this cohort will receive SurgiMend® PRS (ADM) product during the first stage of the reconstruction (expander insertion).
  Other Names: ADM, acellular dermal matrix
  Arms: SurgiMend® PRS (ADM)
Other: No Intervention — Subjects enrolled in to this cohort will not receive an acellular dermal matrix (ADM) product during the first stage of the reconstruction (expander insertion).
  Arms: No Intervention

SUMMARY:
This is a prospective clinical study comparing two-stage breast reconstruction following mastectomy with and without the use of SurgiMend® PRS fetal bovine collagen matrix in patients with pre-mastectomy radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Patient is female
* Patient is undergoing immediate, two-stage breast reconstruction following mastectomy with or without the use of SurgiMend® PRS
* Patient has previously undergone pre-mastectomy XRT for breast cancer, with lumpectomy or partial mastectomy, with the previously irradiated breast now being reconstructed (with or without contralateral mastectomy & reconstruction)
* Patient utilized a textured expander only
* Patient utilized a smooth gel permanent implant only
* Patient has agreed and is able to comply with the study follow-up requirements
* Patient or guardian has provided consent for participation

Exclusion Criteria:

* Patient is undergoing single-stage breast reconstruction
* Patient is undergoing a delayed reconstruction
* Patient is undergoing reconstruction using a smooth tissue expander, textured gel breast implant or any saline breast implant.
* Patient is undergoing planned reconstruction using autologous tissue
* Patient has a known hypersensitivity to collagen or bovine derived materials
* Patient is currently pregnant, nursing, or planning a pregnancy during the course of the study
* Patient who has had pre-mastectomy XRT bilaterally for breast cancer (either at the same time or separated in time)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Capsular Contracture Rate | 12 months Post-Exchange
  Capsular Contracture Rate (Baker III/IV): Reduction from control through 12 months after expander-to-permanent implant exchange
Breast Q | 12 months Post-Exchange
  No decrease in overall patient satisfaction from control as measured by the BREAST-Q Reconstruction Module Patient Satisfaction with Breasts survey, all questions a-p.
  Increase in patient satisfaction from control as measured by the BREAST-Q Reconstruction Module Patient Satisfaction with Breasts survey, questions related to capsular contracture.

SECONDARY OUTCOMES:
No. Capsule Procedures | 12 months Post-Exchange
  Number of capsule procedures performed
Cosmetic Assessment | 12 months Post-Exchange
  Patient: (BREAST-Q Reconstruction Module) Surgeon: (panel review of standard photographs)
Time to Completion | 12 months Post-Exchange
  Time to Completion (expand-to-implant exchange)
Total number of OR procedures | 12 month follow-up visit
  Procedural Attributes: Total number of OR procedures
Total number of visits | 12 month follow up visit
  Procedural Attributes: Total number of ("in office" and OR procedures)